CLINICAL TRIAL: NCT00122551
Title: A Prospective, Randomized, Multicenter Trial of Intermittent Therapy in HIV-Infected Patients With Successful Viral Suppression Under HAART (ANRS 106 Window Trial)
Brief Title: Intermittent Therapy in HIV-1 Infected Patients With Successful Viral Suppression Under Highly Active Antiretroviral Therapy (HAART)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 106 Window
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2005-08-01 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: HIV infections
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: Intermittent antiretroviral therapy

SUMMARY:
Although lifelong continuous therapy with HAART remains the standard of care of HIV infection, allowing to achieve undetectable plasma viral RNA, restore CD4 cell count and provide substantial decline in HIV-related morbidity and mortality, long-term toxicity associated with antiretroviral therapy is a real concern. The purpose of this study is to compare an intermittent therapy strategy to a continuous treatment in patients with chronic and well controlled HIV-1 infection.

DETAILED DESCRIPTION:
Although lifelong continuous therapy with HAART remains the standard of care of HIV infection, allowing to achieve undetectable plasma viral RNA, restore CD4 cell count and provide substantial decline in HIV-related morbidity and mortality, long-term toxicity associated with antiretroviral therapy is a real concern.

The purpose of this study is to compare an intermittent therapy (IT) strategy (8 weeks off / 8 weeks on) to a continuous treatment (CT) in patients with chronic and well controlled HIV-1 infection (CD4 over 450/µl and plasma HIV1-RNA below 200 cp/ml) under HAART, over a 96-week study period.

The study hypothesis is that intermittent therapy is not inferior to continuous therapy in maintaining a CD4 cell above 300/µl. It will compare the proportions of and time to immunological failure (CD4 count below 300/µl confirmed by a retest 14 days later) in the IT and CT groups.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4 cell count over 450/µl for at least 6 months prior to screening
* Plasma HIV1-RNA below 200 cop/ml for at least 6 months prior to screening
* Stable and well tolerated ART for at least 6 months prior to screening
* Acceptable methods of contraception
* Patient able to comply with the protocol
* Informed consent signed prior to (or at) screening

Exclusion Criteria:

* CD4 nadir below 100/µl
* Abacavir or nevirapine in the current ART
* Hepatitis B with 3-TC, adefovir or tenofovir current therapy
* Current or upcoming treatment with interferon for hepatitis B or C
* History of AIDS-defining event in the 18 months prior to screening
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2001-12; Study Completion 2005-04

PRIMARY OUTCOMES:
Immunological failure, defined by a CD4 cell count below 300/µl confirmed by a retest 14 days later during the study

SECONDARY OUTCOMES:
1993 Centers for Disease Control (CDC) classification of HIV infection B or C events
Proportions of patients with CD4 count over 450/µl at week 96
Proportions of patients with plasma HIV load over 400 and 1000/ml thresholds
Plasma and peripheral blood mononuclear cells (PBMC) HIV resistance patterns
Proportions of patients withdrawing initial treatment strategy
Assessment of lipodystrophy and metabolic abnormalities
Antiretroviral therapy (ARTs) adherence assessment
Quality of life assessment
Cost impact of the strategies

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Marchou, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales Hopital Purpan Toulouse; Jean Pierre Aboulker, MD, Study Chair — Inserm SC10
Locations (2):
- France (2):
  - Service des Maladies Infectieuses, Paris
  - Service des Maladies Infectieuses et Tropicales Hopital Purpan, Toulouse

REFERENCES:
- [Derived] Delobel P, Saliou A, Nicot F, Dubois M, Trancart S, Tangre P, Aboulker JP, Taburet AM, Molina JM, Massip P, Marchou B, Izopet J; ANRS 106-Window Study Team. Minor HIV-1 variants with the K103N resistance mutation during intermittent efavirenz-containing antiretroviral therapy and virological failure. PLoS One. 2011;6(6):e21655. doi: 10.1371/journal.pone.0021655. Epub 2011 Jun 27. PMID 21738752
- [Derived] Charreau I, Jeanblanc G, Tangre P, Boyer L, Saouzanet M, Marchou B, Molina JM, Aboulker JP, Durand-Zaleski I; ANRS 106 Study Group. Costs of intermittent versus continuous antiretroviral therapy in patients with controlled HIV infection: a substudy of the ANRS 106 Window Trial. J Acquir Immune Defic Syndr. 2008 Dec 1;49(4):416-21. doi: 10.1097/QAI.0b013e31818a657c. PMID 18931625